CLINICAL TRIAL: NCT02489591
Title: Characterizing Site and Severity of Upper Airway Collapse to Guide Patient Selection for Oral Appliance Therapy for Obstructive Sleep Apnea
Brief Title: Characterizing Upper Airway Collapse to Guide Patient Selection for Oral Appliance Therapy for Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Andrew Wellman, Director, Sleep Disordered Breathing Lab, Brigham and Women's Hospital, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2012P000957
Record Dates: First submitted 2015-06-30; First posted 2015-07-03 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No oral appliance (control) first, oral appliance (BluePro oral appliance or other device) second
- Oral appliance (Experimental): oral appliance (BluePro oral appliance or other device) first, no oral appliance (control) second
  Interventions: Device: Oral appliance; Device: BluePro oral appliance

INTERVENTIONS:
Device: Oral appliance — Patients will bring their prescribed oral appliance.
  Arms: Oral appliance
Device: BluePro oral appliance — Patients without a prescribed oral appliance will have a device provided for the duration of the study (BluePro, BlueSom; used for investigational purposes only). The device provided is a prefabricated thermoplastic customizable mandibular advancement splint.
  Arms: Oral appliance

SUMMARY:
Obstructive Sleep Apnea (OSA) is characterized by collapse of one or more pharyngeal structures during sleep (velum, tongue base, lateral walls, epiglottis). Structure-specific therapies for OSA have emerged as alternatives to positive airway pressure (PAP). Oral appliance (OA) therapy is increasingly being indicated for OSA treatment, although a complete response occurs in approximately 50% of patients. In general, OA devices are designed to maintain the mandible and/or tongue in a protruded posture during sleep, preventing upper airway obstruction. Limited studies in awake or sedated patients have demonstrated the effects of mandibular advancement on aspects of pharyngeal structure and function. The objective of the proposed research is to fully characterize upper airway collapse in OSA patients during natural sleep and use this information to understand why some patients appear to exhibit a large improvement in pharyngeal collapsibility whereas others do not.

DETAILED DESCRIPTION:
OSA patients will undergo a baseline sleep endoscopy study to identify the site of pharyngeal collapse. Subsequently, they will undergo two clinical polysomnographies (PSGs) to measure the effect of an oral appliance (a site specific therapy) on upper airway collapsibility and sleep apnea severity. During the first hour of each clinical PSG, the passive pharyngeal collapsibility will be determined using the standard 5-breath continuous positive airway pressure (CPAP) drop method. During the remainder of the night, patients will be monitored to determine sleep apnea severity (apnea-hypopnea index). These measurements will allow the investigators to determine which pharyngeal collapsing site responds best (both in terms of collapsibility and AHI) to mandibular advancement with an oral appliance. Patients who have their own oral appliance will be recruited. In addition, patients without an oral appliance will be provided with a temporary oral appliance for the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Obstructive Sleep Apnea

Exclusion Criteria:

* Any unstable cardiac condition (other than well controlled hypertension) or pulmonary problems.
* Any medication known to influence breathing, sleep/arousal or muscle physiology
* Concurrent sleep disorders (insomnia, narcolepsy, central sleep apnea or parasomnia)
* Claustrophobia
* Inability to sleep supine
* Periodontal disease and/or insufficient number of teeth
* Allergy to lidocaine or oxymetazoline hydrochloride
* For women: Pregnancy

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-07-14 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Change in passive pharyngeal collapsibility (OA therapy minus control) | 3 nights
  The passive pressure-flow relationship is characterized by the critical closing pressure (Pcrit) , and the ventilatory flow at atmospheric pressure ( V passive). Pcrit and V passive will be determined using the standard 5-breath CPAP drop method.
  The change in collapsibility will be compared across subgroups defined by the site of collapse measured using sleep-endoscopy. Patients will sleep supine for this measurement.
Change in sleep apnea severity (AHI) | 2 nights
  The change in apnea-hypopnea index (AHI, 3% desaturation or arousal criteria; OA therapy minus control) will be compared across subgroups defined by the site of collapse measured using sleep-endoscopy. Baseline collapsibility will be incorporated as a predictor of the change in AHI.

SECONDARY OUTCOMES:
Change in peak flow during sleep (OA therapy minus control) | 2 nights
  During the portion of the night dedicated to measuring sleep apnea severity, peak flow will also be measured during sleep to quantify activated upper airway collapsibility.
Objective sleep quality (OA therapy minus control) | 2 nights
  Arousal index, one of the standard measures of sleep quality, will be assessed.
Objective sleep quality (OA therapy minus control) | 2 nights
  Proportion of sleep in Non rapid eyes movement ( NREM) stage 1,one of the standard measures of sleep quality, will be assessed.
Subjective sleep quality (OA therapy minus control) | 2 nights
  Patients will rate whether they slept better/worse/same with the OA vs control.

CONTACTS AND LOCATIONS:
Overall Officials: David A Wellman, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States